CLINICAL TRIAL: NCT00605891
Title: A Randomized, Controlled,14-Treatment Day, Multicenter Study to Determine the Optimal Efficacious and Safe Dose of CHF 4226 in a Metered Dose Inhaler in Treating Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Dose Finding Study of CHF 4226 for Treating Patients With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Collaborators: Chiesi USA, Inc. (Industry)
Responsible Party: Steven Linberg/ Managing Director, Chiesi Pharmaceuticals Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: US/PR/033009/001/05; EudraCT Number: 2006-000531-10
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — carmoterol; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- A (Experimental): carmoterol (CHF 4226) 1.0 μg once a day, in the morning
  Interventions: Drug: carmoterol (CHF 4226)
- B (Experimental): carmoterol (CHF 4226) 2.0 μg once a day, in the morning
  Interventions: Drug: carmoterol (CHF 4226)
- C (Experimental): carmoterol (CHF 4226) 4.0 μg once a day, in the morning
  Interventions: Drug: carmoterol (CHF 4226)
- D (Placebo Comparator): Placebo once a day, in the morning
  Interventions: Drug: placebo
- E (Active Comparator): Salmeterol 50 μg BID, in the morning and in the evening
  Interventions: Drug: salmeterol

INTERVENTIONS:
Drug: carmoterol (CHF 4226) — carmoterol pMDI 2.0 μg once a day, in the morning
  (1 puff of carmoterol 1.0 mcg + 1 puff of carmoterol 1.0 mcg)
  Other Names: CHF 4226
  Arms: B
Drug: carmoterol (CHF 4226) — carmoterol pMDI 1.0 μg once a day, in the morning
  (1 puff of carmoterol 1.0 mcg + 1 puff of placebo pMDI))
  Other Names: CHF 4226
  Arms: A
Drug: carmoterol (CHF 4226) — carmoterol pMDI 4.0 μg once a day, in the morning
  (1 puff of carmoterol 2.0 mcg + 1 puff of carmoterol 2.0 mcg)
  Other Names: CHF 4226
  Arms: C
Drug: salmeterol — Salmeterol 50 μg DPI, in the morning and in the evening (1 blister BID)
  Other Names: Serevent® Diskus®/Accuhaler®
  Arms: E
Drug: placebo — Placebo pMDI once a day, in the morning (1 puff of placebo pMDI + 1 puff of placebo pMDI)
  Arms: D

SUMMARY:
The purpose of this study is to identify the optimal once-daily dose of CHF 4226 to be further developed for the treatment of patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed an IRB-/Ethics Committee-approved Informed Consent form
* Patient is a male or non-pregnant female between the ages of 40 - 75 years, inclusive
* Patient has a current or past smoking history of at least 15 pack-years
* Patient has a clinical diagnosis of COPD in accordance with the recommendations of the National Heart Lung and Blood Institute/World Health Organization (NHLBI/WHO) Global Initiative for Chronic Obstructive Lung Disease (GOLD)
* Patient meets the following requirements after an FEV1 albuterol reversibility test (i.e., 30 minutes following 200 mcg (metered dose) albuterol/salbutamol pMDI):
* FEV1 is at least 0.9L
* FEV1 of 40% - 70%, inclusive, of patient's predicted normal value
* Change in FEV1 > 4% of patient's predicted normal value

  * If change in FEV1 < 4% of patient's predicted normal value, then this requirement must be met after retesting during the run-in period, at least 24 hours prior to Day -1
* FEV1/FVC < 70%

Exclusion Criteria:

* Patient has a history of asthma, allergic rhinitis, or atopy
* Patient has a blood eosinophil count > 500/microliter
* Patient had a COPD exacerbation or a lower respiratory tract infection within 8 weeks prior to screening, or during the run-in period, that resulted in the use of an antibiotic, or oral or parenteral corticosteroids
* Patient is on an inhaled corticosteroid that has been initiated, or the effective dose has been changed, within 4 weeks prior to screening or during the run-in period
* Patient has an uncontrolled cardiovascular (e.g., uncontrolled hypertension), respiratory, hematologic, immunologic, renal, neurologic, hepatic, endocrine (e.g., uncontrolled diabetes mellitus) or other disease, or any condition that might, in the judgment of the Investigator, place the patient at undue risk or potentially compromise the results or interpretation of the study
* Patient has a history of coronary artery disease, cerebrovascular disease, cardiac arrhythmias
* Patient has a concomitant disease of poor prognosis (e.g., cancer)
* Patient has a serum potassium value ≤ 3.5 mEq/L or >5.5mEq/L and/or a fasting serum glucose value ≥ 140 mg/dL
* Patient has an abnormal QTc Fridericia interval value in the Screening visit ECG test (i.e., > 450 msec in males or > 470 msec in females)
* Patient has developed Cor Pulmonale
* Patient is receiving long term oxygen therapy, i.e., ≥ 16 hours/24-hour period, every day
* Patient has a known intolerance/hypersensitivity to Beta2-adrenergic agonists, propellant gases/excipients
* Patient is receiving treatment with a tricyclic antidepressant or a monoamine oxidase inhibitor (MAOI)
* Patient has received a live-attenuated virus vaccination within two weeks prior to screening or during the run-in
* Patient is pregnant or lactating female, or female at risk of pregnancy (i.e., not using an adequate contraceptive method)
* Patient is mentally or legally incapacitated
* Patient has participated in another investigational study within 30 days prior to screening
* Patient abuses alcohol or other substances
* Patient is potentially non-compliant or unable to perform required outcome measurements of the protocol

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2006-10; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 | Day 1 to Day 14 (+3 days)

SECONDARY OUTCOMES:
FEV1 | 10 and 30 min, 1, 2, and 3 hrs post dose on Day 1, Day 2 and Day 14 (+3)
ECG/QTc | pre dose and post dose at 30' on Days 1, 2 and 14 (+3)
Fasting serum potassium | pre dose and post dose at 30' on Days 1, 2 and 14 (+3)
Fasting glucose | pre dose and post dose at 30' on Days 1, 2 and 14 (+3)
Change in FEV1 | 10 and 30 min, 1, 2, and 3 hrs post dose on Day 1, Day 2 and Day 14 (+3)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Make, MD, Principal Investigator — National Jewish Medical & Research Center; Steven E Linberg, Ph.D., Study Director — Chiesi Farmaceutici S.p.A.
Locations (50):
- United States (24):
  - Clopton Clinic, Jonesboro, Arkansas
  - ABM Research Center, Fresno, California
  - UCSD - Clinical Trials Center, San Diego, California
  - Institute of Healthcare Assessment Inc., San Diego, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Clinical Research of West Florida, Clearwater, Florida
  - University Clinical Research - DeLand, LLC, DeLand, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Edward Hospital and Helath Services, Center for Clinical Trials, Naperville, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - ClinSite, LLC, Ann Arbor, Michigan
  - ClinSite, Canton, Michigan
  - Delaware Valley Clinical Research, Cherry Hill, New Jersey
  - Carolina Pharmaceutical Research, Statesville, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - Clinical Research Institute of Southern Oregon PC, Medford, Oregon
  - Pulmonary Consultants - Research Department, Medford, Oregon
  - Lowcountry Lung and Critical Care, PA, North Charleston, South Carolina
  - Amarillo Center for Clinical Research, Ltd., Amarillo, Texas
  - Breath of Life Research Institute, Katy, Texas
  - The University of Texas Health Center at Tyler, Tyler, Texas
  - University of Wisconsin-Allergy/Asthma, Madison, Wisconsin
- Czechia (7):
  - Ordinace pro nemoci dychaciho ustroji, Beroun
  - OTRAN, Kutná Hora
  - Plicni a alergologicka ambulance, Kutná Hora
  - Pneumolog, internista, Lovosice
  - Nemocnice Na Homolce Plicni ambulance, Prague
  - Plicni ambulance, Praha 3 - Zizkov
  - Plicni ambulance Rokycany, Rokycany
- Germany (7):
  - Medars GmbH, Berlin
  - Lungenzentrum Geesthacht, Geesthacht
  - Pneumologisches Forschungsinstitut GmbH, Großhansdorf
  - Pneumologisches Forschungsinstitut Niederlassung Hamburg, Hamburg
  - Robert-Koch-Klinik, Leipzig
  - SMO, MD GmbH, Magdeburg
  - IFG GmbH, Rüdersdorf
- Poland (4):
  - Medcare Specjalistyczna Opieka Medyczna NZOZ, Gdansk
  - NZOZ Non-nocere, Gdansk
  - Klinika Pulmonologii i Alergologii, Lodz
  - SPZOZ w Proszowicach Oddzial Chorob Pluc, Proszowice
- Romania (6):
  - Spitalul Clinic Judetean de Urgenta Brasov, Brasov
  - Spitalul de Urgenta "Prof. Dr. Dimitrie Gerota", Bucharest
  - Spitalul Clinic de Urgenta Militar Central "Davila", Bucharest
  - Spitalul Clinic "Sf. Maria", Bucharest
  - Institutul National de Pneumoftisiologie "M. Nasta", Bucharest
  - Spitalul de Pneumoftiziologie Constanta, Constanța
- South Africa (2):
  - UCT Lung Institute, Mowbray, Cape Town
  - Tiervlei Trial Center, Karl Bremer Hospital, Bellville

REFERENCES:
- [Background] Matera MG, Cazzola M. ultra-long-acting beta2-adrenoceptor agonists: an emerging therapeutic option for asthma and COPD? Drugs. 2007;67(4):503-15. doi: 10.2165/00003495-200767040-00002. PMID 17352511
- [Background] Cazzola M, Matera MG, Lotvall J. Ultra long-acting beta 2-agonists in development for asthma and chronic obstructive pulmonary disease. Expert Opin Investig Drugs. 2005 Jul;14(7):775-83. doi: 10.1517/13543784.14.7.775. PMID 16022567
- [Background] Matsukawa M, Takeda K, Shima H, Tagawa K, Banno K, Sato T. Enzyme-linked immunosorbent assay for TA-2005-glucuronide in human plasma. J Pharm Biomed Anal. 1998 Jun;17(2):245-54. doi: 10.1016/s0731-7085(97)00186-6. PMID 9638577
- [Background] Kikkawa H, Isogaya M, Nagao T, Kurose H. The role of the seventh transmembrane region in high affinity binding of a beta 2-selective agonist TA-2005. Mol Pharmacol. 1998 Jan;53(1):128-34. doi: 10.1124/mol.53.1.128. PMID 9443940
- [Background] Rossoni G, Manfredi B, Razzetti R, Civelli M, Bongrani S, Berti F. Positive interaction of the beta2-agonist CHF 4226.01 with budesonide in the control of bronchoconstriction induced by acetaldehyde in the guinea-pigs. Br J Pharmacol. 2005 Feb;144(3):422-9. doi: 10.1038/sj.bjp.0706096. PMID 15655502
- [Background] Rossoni G, Manfredi B, Razzetti R, Civelli M, Berti F. Positive interaction of the novel beta2-agonist carmoterol and tiotropium bromide in the control of airway changes induced by different challenges in guinea-pigs. Pulm Pharmacol Ther. 2007;20(3):250-7. doi: 10.1016/j.pupt.2006.01.004. Epub 2006 Mar 14. PMID 16533614
- [Background] Voss HP, Shukrula S, Wu TS, Donnell D, Bast A. A functional beta-2 adrenoceptor-mediated chronotropic response in isolated guinea pig heart tissue: selectivity of the potent beta-2 adrenoceptor agonist TA 2005. J Pharmacol Exp Ther. 1994 Oct;271(1):386-9. PMID 7965739
- [Background] Kikkawa H, Kanno K, Ikezawa K. TA-2005, a novel, long-acting, and selective beta 2-adrenoceptor agonist: characterization of its in vivo bronchodilating action in guinea pigs and cats in comparison with other beta 2-agonists. Biol Pharm Bull. 1994 Aug;17(8):1047-52. doi: 10.1248/bpb.17.1047. PMID 7820105
- [Background] Voss HP, Donnell D, Bast A. Atypical molecular pharmacology of a new long-acting beta 2-adrenoceptor agonist, TA 2005. Eur J Pharmacol. 1992 Dec 1;227(4):403-9. doi: 10.1016/0922-4106(92)90158-r. PMID 1359974
- [Background] Kikkawa H, Naito K, Ikezawa K. Tracheal relaxing effects and beta 2-selectivity of TA-2005, a newly developed bronchodilating agent, in isolated guinea pig tissues. Jpn J Pharmacol. 1991 Oct;57(2):175-85. doi: 10.1254/jjp.57.175. PMID 1687479
- [Background] Spadari-Bartfisch RC, Santos IN, Vanderlei LC, Marcondes FK. Pharmacological evidence for beta2-adrenoceptor in right atria from stressed female rats. Can J Physiol Pharmacol. 1999 Jun;77(6):432-40. PMID 10537229
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2006-000531-10